CLINICAL TRIAL: NCT00634985
Title: A Multicentre, Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of Eletriptan 40 Mg for the Treatment of Migraine (With or Without Aura) in Subjects Unsuccessfully Treated With NSAIDS
Brief Title: Safety and Efficacy of Eletriptan for the Treatment of Migraine in Subjects Unsuccessfully Treated With Nonsteroidal Anti-inflammatory Drugs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1601085
Record Dates: First submitted 2008-03-03; First posted 2008-03-13 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — eletriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: eletriptan

INTERVENTIONS:
Drug: eletriptan — 40 mg oral tablet for migraine attack; additional 40 mg oral tablet >2 hours from first dose if migraine reoccurred within 24 hours of achieving response

SUMMARY:
To assess the safety and efficacy of eletriptan for the treatment of migraine in subjects who had not been adequately treated with non-steroidal antiinflammatory drugs (NSAIDs)

ELIGIBILITY:
Inclusion Criteria:

* Met International Headache Society diagnostic criteria for migraine with or without aura
* Expected to suffer one to six acute migraine attacks per month based on past history
* Experienced migraines for at least one year prior to entering study, and historically have not responded to NSAIDs

Exclusion Criteria:

* Frequent migraine or frequent concomitant non-migrainous headache (average of >6 attacks per month)
* Atypical migraines that consistently failed to respond to adequate medical therapy
* Migraine with prolonged aura, familial hemiplegic migraine, basilar migraine, migrainous infarction, migraine aura without headache, or migraine with acute-onset aura

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2002-11; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Headache severity and response post-treatment | 2 hours
Functional response post-treatment | 2 hours

SECONDARY OUTCOMES:
Presence of associated symptoms including, nausea, vomiting, phonophobia, and photophobia at baseline and post-treatment | 1, 2, 4, and 24 hours
Migraine recurrence post-treatment | 1, 2, 4, and 24 hours
Time loss (from normal activities and from work) post-treatment | 24 hours
Subject preference and acceptability post-treatment | 24 hours and 12 weeks
Subject satisfaction post-treatment | 2 and 24 hours
Adverse events | Week 12
Physical examination | Week 12
Vital signs | Week 12
Electrocardiogram | Week 12
Headache severity and response at baseline and post-treatment | 1, 4 and 24 hours
Functional impairment severity and response at baseline and post-treatment | 1, 4 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Turkey (Türkiye) (5):
  - Pfizer Investigational Site, Çapa, Istanbul
  - Pfizer Investigational Site, Gaziantep
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Izmir
  - Pfizer Investigational Site, Samsun
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1601085&StudyName=Safety%20and%20Efficacy%20of%20Eletriptan%20for%20the%20Treatment%20of%20Migraine%20in%20Subjects%20Unsuccessfuly%20Treated%20with%20Nonsteroidal%20Anti-inflammatory%20Drugs